CLINICAL TRIAL: NCT04203446
Title: Assessment of Clinical Factors Influencing on Correctness of Inhalation Technique in Adults With Asthma or COPD.
Brief Title: Factors Influencing on Correctness of Inhalation Technique.
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, Principal Investigator, Medical University of Warsaw
Other Study IDs: Inhalation technique 1
Record Dates: First submitted 2019-08-24; First posted 2019-12-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Asthma; COPD
Keywords: inhalation technique
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with asthma or COPD: Adults (18-85 years old) with asthma or COPD diagnosed at least 3 months earlier, who are regularly treated with at least one inhlaer daily
  Interventions: Other: Assessment of correctness of inhaling technique

INTERVENTIONS:
Other: Assessment of correctness of inhaling technique — Assessment of correctness of inhaling technique in patients with asthma or COPD

SUMMARY:
Asthma and COPD are common chronic diseases of respiratory system. The correct use of inhalers is crucial in terms of efficacy of the treatment, however both asthma and COPD patients quite frequently misuse the inhalers. The objective of this study is to determine the factors influencing the number of inhalation errors committed by asthma and COPD patients when using the inhalers.

In included patients the inhalation technique will be evaluated (by both list of inhalation errors and 4 point scale of proper inhaling) by two observers and the below information will be collected:

* general demographic information and education level
* information concerning time of diagnosis, the previous course of disease, smoking history, number of previous inhalation techniques training, the sources of information about the inhalation technique and adherence to therapy
* Asthma Control Test or COPD Assessment Test (respectively for asthma and COPD)
* assessment of quality of life (St. George's Questionnaire for COPD and Asthma Quality of Life Questionnaire for asthma)
* cognitive functions assessment using Mini-Mental State Examination
* the simplified assessment of vision impairments
* the results of spirometry

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are common chronic diseases of respiratory system. Asthma affects about 5% of adults in Poland. The inhaling therapy is the cornerstone of asthma treatment, especially inhaled glucocorticosteroids (ICS). The correct use of inhalers is crucial for efficiency of the therapy and reduction of undesirable side effects of medications. COPD is also a common chronic respiratory disease that affects about 10% of adults above 40 years old. The most important action to prevent and to treat COPD is to stop smoking. The main medications used by COPD patients are inhaled bronchodilators. Both asthma and COPD patients misuse the inhalers.

The objective of this study is to determine the factors influencing the number of inhalation errors committed by asthma and COPD patients when using the inhalers.

Patients:

Patients with asthma or COPD treated in hospital or in out-patient clinic will be asked for participating in the study. Power analysis and sample size calculations indicated that a sample size of 215 subjects (with either asthma or COPD) would provide statistical power to detect even weak correlation (r=0.2) assuming error alpha = 0.05, beta = 0.20 and 10% drop out.

Study design

In included patients inhalation technique will be evaluated (by both list of inhalation errors and 4 point scale of proper inhaling) by two observers and the below information will be gathered:

* general demographic information and education level
* information concerning time of diagnosis, the previous course of disease, smoking history, number of previous inhalation techniques training, the sources of information about the inhalation technique and adherence to therapy
* Asthma Control Test and COPD Assessment Test respectively for asthma and COPD
* assessment of quality of life with the disease (St. George's Questionnaire for COPD and Asthma Quality of Life Questionnaire for asthma)
* cognitive functions assessment using Mini-Mental State Examination
* the simplified assessment of vision impairments
* the results of spirometry The main outcome will be correlation between inhalation technique and other above mentioned factors.

Identification of factors influencing the inhaling errors in patients with asthma or COPD will enable to plan the actions to improve the efficiency of inhaler medications use. At the end of the study all patients will be taught how to use their inhalers properly.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent for participating in the study
2. Age 18 -85 years
3. COPD or asthma diagnosed at least 3 months prior to enrolment
4. using of at least one inhaler regularly every day
5. using one of the inhalers: Metered Dose Inhalers (MDI), Dry Powder Inhalers (DPI) or Metered Dose Liquid Inhalers (MDLI)

Exclusion Criteria:

1. Lack of informed consent
2. Age <18 years or > 85 years old
3. Diagnosis of asthma or COPD shorter than 3 months before enrollment
4. Using inhalers unregularly.
5. Symptoms of infection 5 days prior to beginning of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with asthma or COPD treated in hospital or in out-patient clinic will be asked for participating in the study
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Assessment of correctness of inhalation technique | baseline
  Assessment of correctness of inhalation technique by list of inhalation errors and 4 point scale of proper inhaling and by two observers

SECONDARY OUTCOMES:
Assessment of general demographic features | baseline
  age (years)
Assessment of educational level | baseline
  educational level (basic, secondary, higher)
Assessment of general demographic features | baseline
  smoking history (pack/years)
Assessment of asthma or COPD duration | baseline
  asthma or COPD duration
Assessment of asthma or COPD severity | baseline
  Asthma Control Test score or COPD Assessment Test score respectively for asthma and COPD
Assessment of quality of life related to COPD | baseline
  St. George's Questionnaire score for COPD
Assessment of quality of life related to asthma | baseline
  Asthma Quality of Life Questionnaire score for asthma
Assessment of earlier training in inhalation technique | baseline
  number of earlier trainings in inhalation technique
Assessment of patient's adherence | baseline
  number of days with missed doses of inhaled drugs per month
Assesment of basic cognitive function | baseline
  Mini-Mental State Examination score
Assessment of vision impairments | baseline
  assessment of vision impairments by Snellen vision test boards

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Krenke, MD,PhD,Prof, Study Director — Warsaw Medical Univeristy
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Result] Laube BL, Janssens HM, de Jongh FH, Devadason SG, Dhand R, Diot P, Everard ML, Horvath I, Navalesi P, Voshaar T, Chrystyn H; European Respiratory Society; International Society for Aerosols in Medicine. What the pulmonary specialist should know about the new inhalation therapies. Eur Respir J. 2011 Jun;37(6):1308-31. doi: 10.1183/09031936.00166410. Epub 2011 Feb 10. PMID 21310878
- [Result] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Result] Normansell R, Kew KM, Mathioudakis AG. Interventions to improve inhaler technique for people with asthma. Cochrane Database Syst Rev. 2017 Mar 13;3(3):CD012286. doi: 10.1002/14651858.CD012286.pub2. PMID 28288272
- [Result] Sanchis J, Gich I, Pedersen S; Aerosol Drug Management Improvement Team (ADMIT). Systematic Review of Errors in Inhaler Use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406. doi: 10.1016/j.chest.2016.03.041. Epub 2016 Apr 7. PMID 27060726
- [Result] Usmani OS, Lavorini F, Marshall J, Dunlop WCN, Heron L, Farrington E, Dekhuijzen R. Critical inhaler errors in asthma and COPD: a systematic review of impact on health outcomes. Respir Res. 2018 Jan 16;19(1):10. doi: 10.1186/s12931-017-0710-y. PMID 29338792